CLINICAL TRIAL: NCT00312806
Title: Real Life: Treatment Response in Patients With Symptoms Due to Gastroesophageal Reflux Disease Either With or Without Esophagitis Treated With Pantoprazole Sodium 40 mg o.d. Over 8 Weeks
Brief Title: Effect of Pantoprazole on the Symptoms of Acid Reflux Disease in Adult Patients (BY1023/M3-341)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/M3-341
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease; GERD; Pantoprazole; ReQuestTM
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole 40 mg o.d.

SUMMARY:
The aim of the present study is to identify factors (such as symptom patterns and symptom scores) that influence the response to treatment with pantoprazole using different evaluation methods (e.g., ReQuest™ questionnaire, patient and investigator assessment). Pantoprazole will be administered once daily in the morning at one dose level. The study duration consists of a treatment period of 8 weeks. The study will provide further data on safety and tolerability of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Outpatients of at least 18 years (21 years in Argentina)
* Patient considered to have GERD symptoms

Main Exclusion Criteria:

* Acute peptic ulcer and/or ulcer complications
* Systemic glucocorticoids or non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2-inhibitors (> 5 days on demand but not more than 3 consecutive days) during the last 28 days before study start (except regular intake of acetylsalicylic acid at a dose up to 163 mg/day)
* Intake of proton pump inhibitors during the last 10 days before study start
* Female patients of childbearing potential not using adequate means of birth control
* Pregnant or breast-feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Response to treatment with pantoprazole at week 8, as measured by the questionnaire ReQuest™ | 8 weeks

SECONDARY OUTCOMES:
Response to treatment with pantoprazole at week 4, as measured by the questionnaire ReQuest™ | 4 and 8 weeks
Investigator assessment | 4 and 8 weeks
Safety and efficacy | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Ulmer, MD, Principal Investigator — Medical practice, D-71640 Ludwigsburg, Germany
Locations (157):
- Argentina (2):
  - Altana Pharma/Nycomed, Buenos Aires
  - Altana Pharma/Nycomed, La Plata
- Australia (10):
  - Altana Pharma/Nycomed, Bedford Park SA
  - Altana Pharma/Nycomed, Bondi Junction
  - Altana Pharma/Nycomed, Fitzroy
  - Altana Pharma/Nycomed, Footscray
  - Altana Pharma/Nycomed, Fremantle, WA
  - Altana Pharma/Nycomed, Kippa_ring
  - Altana Pharma/Nycomed, Melbourne
  - Altana Pharma/Nycomed, NSW
  - Altana Pharma/Nycomed, Penrith, NSW
  - Altana Pharma/Nycomed, Phrahran
- Austria (7):
  - Altana Pharma/Nycomed, Deutschlandsberg
  - Altana Pharma/Nycomed, Feldbach
  - Altana Pharma/Nycomed, Graz
  - Altana Pharma/Nycomed, Krems A. D. Donau
  - Altana Pharma/Nycomed, Lilienfeld
  - Altana Pharma/Nycomed, Sankt Pölten
  - Altana Pharma/Nycomed, Vienna
- Belgium (12):
  - Altana Pharma/Nycomed, Bouge
  - Altana Pharma/Nycomed, Brussels
  - Altana Pharma/Nycomed, Edegem
  - Altana Pharma/Nycomed, Eupen
  - Altana Pharma/Nycomed, Ghent
  - Altana Pharma/Nycomed, Jette
  - Altana Pharma/Nycomed, Kortrijk
  - Altana Pharma/Nycomed, Leuven
  - Altana Pharma/Nycomed, Merksem
  - Altana Pharma/Nycomed, Ostend
  - Altana Pharma/Nycomed, Saint Niklaas
  - Altana Pharma/Nycomed, Sart-Tilman/Liege 1
- Brazil (11):
  - Altana Pharma/Nycomed, Belo Horizonte - Minas Gerais
  - Altana Pharma/Nycomed, Botucatu - SP CEP
  - Altana Pharma/Nycomed, Campinas - Sao Paulo
  - Altana Pharma/Nycomed, Campinas /SP
  - Altana Pharma/Nycomed, Curitiba-PR
  - Altana Pharma/Nycomed, Ilha Do Fundao - Rio de Janeiro - RJ
  - Altana Pharma/Nycomed, Pinheiros Sao Paulo - SP
  - Altana Pharma/Nycomed, Porto Alegre
  - Altana Pharma/Nycomed, Porto Alegre - RS
  - Altana Pharma/Nycomed, Porto Alegre-RS
  - Altana Pharma/Nycomed, Ribeirao Preto-SP
- Canada (12):
  - Altana Pharma/Nycomed, Abbotsford, BC
  - Altana Pharma/Nycomed, Calgary
  - Altana Pharma/Nycomed, Hamilton
  - Altana Pharma/Nycomed, London
  - Altana Pharma/Nycomed, Montreal
  - Altana Pharma/Nycomed, Montreal, QC
  - Altana Pharma/Nycomed, Québec
  - Altana Pharma/Nycomed, St.-Charles Borromee, QC
  - Altana Pharma/Nycomed, Ste Foy
  - Altana Pharma/Nycomed, Toronto
  - Altana Pharma/Nycomed, Windsor
  - Altana Pharma/Nycomed, Winnipeg
- France (12):
  - Altana Pharma/Nycomed, Agen
  - Altana Pharma/Nycomed, Bobigny
  - Altana Pharma/Nycomed, Hagondange
  - Altana Pharma/Nycomed, Joué-lès-Tours
  - Altana Pharma/Nycomed, Lamballe
  - Altana Pharma/Nycomed, Marseille
  - Altana Pharma/Nycomed, Metz
  - Altana Pharma/Nycomed, Orthez
  - Altana Pharma/Nycomed, Saint-Mandé
  - Altana Pharma/Nycomed, Toul
  - Altana Pharma/Nycomed, Toulouse
  - Altana Pharma/Nycomed, Troyes
- Germany (9):
  - Altana Pharma/Nycomed, Bonn
  - Altana Pharma/Nycomed, Burg
  - Altana Pharma/Nycomed, Gardelegen
  - Altana Pharma/Nycomed, Heilbronn
  - Altana Pharma/Nycomed, Hennef (Sieg)
  - Altana Pharma/Nycomed, Ludwigsburg
  - Altana Pharma/Nycomed, Lübeck
  - Altana Pharma/Nycomed, Magdeburg
  - Altana Pharma/Nycomed, Schwerin
- Altana Pharma/Nycomed, Hong Kong, Hong Kong
- India (8):
  - Altana Pharma/Nycomed, Coimbatore
  - Altana Pharma/Nycomed, Hyderabad
  - Altana Pharma/Nycomed, Jaipur
  - Altana Pharma/Nycomed, Madurai
  - Altana Pharma/Nycomed, Mumbai
  - Altana Pharma/Nycomed, Mysore
  - Altana Pharma/Nycomed, Nagpur
  - Altana Pharma/Nycomed, Pune
- Italy (11):
  - Altana Pharma/Nycomed, Aviano (Pordenone)
  - Altana Pharma/Nycomed, Bari
  - Altana Pharma/Nycomed, Caserta
  - Altana Pharma/Nycomed, Catania
  - Altana Pharma/Nycomed, Genova
  - Altana Pharma/Nycomed, Mestre (VE)
  - Altana Pharma/Nycomed, Milan
  - Altana Pharma/Nycomed, Napoli
  - Altana Pharma/Nycomed, Parma
  - Altana Pharma/Nycomed, Roma
  - Altana Pharma/Nycomed, Rozzano (Milano)
- Malaysia (2):
  - Altana Pharma/Nycomed, Kota Kinabalu, Sabah
  - Altana Pharma/Nycomed, Kuala Lumpur
- Mexico (10):
  - Altana Pharma/Nycomed, Col Del Valle, México D.F.
  - Altana Pharma/Nycomed, Col Héroes de Padierna, México D.F.
  - Altana Pharma/Nycomed, Col. Altavista,Tampico Tamaulipas,Mexico
  - Altana Pharma/Nycomed, Col. Ex Hacienda Coapa Mexico D.F.
  - Altana Pharma/Nycomed, Héroes de Padierna, México D.F.
  - Altana Pharma/Nycomed, León, Guanajuato Mexico
  - Altana Pharma/Nycomed, León, Guanajuato
  - Altana Pharma/Nycomed, Lomas de Chapultepec, México D.F.
  - Altana Pharma/Nycomed, México, D.F.
  - Altana Pharma/Nycomed, Villahermosa, Tabasco
- Poland (4):
  - Altana Pharma/Nycomed, Bialystok
  - Altana Pharma/Nycomed, Katowice
  - Altana Pharma/Nycomed, Lodz
  - Altana Pharma/Nycomed, Warsaw
- Portugal (8):
  - Altana Pharma/Nycomed, Amadora
  - Altana Pharma/Nycomed, Carnaxide
  - Altana Pharma/Nycomed, Coimbra
  - Altana Pharma/Nycomed, Lisbon
  - Altana Pharma/Nycomed, Santarém
  - Altana Pharma/Nycomed, Setúbal
  - Altana Pharma/Nycomed, Viana do Castelo
  - Altana Pharma/Nycomed, Vila Nova de Gaia
- Altana Pharma/Nycomed, Singapore, Singapore
- South Africa (8):
  - Altana Pharma/Nycomed, Berea, Durban
  - Altana Pharma/Nycomed, Bloemfontein
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, eManzimtoti
  - Altana Pharma/Nycomed, Panorama
  - Altana Pharma/Nycomed, Port Elizabeth
  - Altana Pharma/Nycomed, Pretoria
  - Altana Pharma/Nycomed, Somerset West
- Altana Pharma/Nycomed, Seoul, South Korea
- Spain (9):
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, Cadiz
  - Altana Pharma/Nycomed, Castellon
  - Altana Pharma/Nycomed, Córdoba
  - Altana Pharma/Nycomed, Granada
  - Altana Pharma/Nycomed, Madrid
  - Altana Pharma/Nycomed, Pamplona
  - Altana Pharma/Nycomed, Ribeira
  - Altana Pharma/Nycomed, Seville
- Switzerland (10):
  - Altana Pharma/Nycomed, Basel
  - Altana Pharma/Nycomed, Biasca
  - Altana Pharma/Nycomed, Biel/Bienne
  - Altana Pharma/Nycomed, Lausanne 11 VD
  - Altana Pharma/Nycomed, Liestal
  - Altana Pharma/Nycomed, Locarno, TI.
  - Altana Pharma/Nycomed, Lucerne
  - Altana Pharma/Nycomed, Payerne
  - Altana Pharma/Nycomed, Thun
  - Altana Pharma/Nycomed, Zurich
- Taiwan (3):
  - Altana Pharma/Nycomed, Taichung
  - Altana Pharma/Nycomed, Tainan
  - Altana Pharma/Nycomed, Taipei
- United Kingdom (6):
  - Altana Pharma/Nycomed, Bath
  - Altana Pharma/Nycomed, Blackpool
  - Altana Pharma/Nycomed, Glasgow
  - Altana Pharma/Nycomed, Middlesex
  - Altana Pharma/Nycomed, Sheffield
  - Altana Pharma/Nycomed, Trowbridge

REFERENCES:
- [Derived] Goh KL, Choi KD, Choi MG, Hsieh TY, Jung HY, Lien HC, Menon J, Mesenas S, Park H, Sheu BS, Wu JC. Factors influencing treatment outcome in patients with gastroesophageal reflux disease: outcome of a prospective pragmatic trial in Asian patients. BMC Gastroenterol. 2014 Sep 9;14:156. doi: 10.1186/1471-230X-14-156. PMID 25200403
- [Derived] Heading RC, Monnikes H, Tholen A, Schmitt H. Prediction of response to PPI therapy and factors influencing treatment outcome in patients with GORD: a prospective pragmatic trial using pantoprazole. BMC Gastroenterol. 2011 May 11;11:52. doi: 10.1186/1471-230X-11-52. PMID 21569313